CLINICAL TRIAL: NCT04480008
Title: Resilient Living Program for Patients With Advanced Cancer and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deirdre R. Pachman, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-011510; NCI-2021-02776 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2020-07-02; First posted 2020-07-21 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resilient Living Program (Experimental): All participants will be in the Resilient Living Program arm. Study participation involves participating in a 12-week stress management and resilience training program. This will involve four virtual sessions (video or phone) and answering questions about their health, well-being, and quality of life. There will also be online modules to watch and an accompanying journal (with prompts) to keep.
  Interventions: Behavioral: Resilient Living Program

INTERVENTIONS:
Behavioral: Resilient Living Program — Participants will be given the journal Resilient Living with Dr. Sood: Building Strength for Difficult Days to use throughout the study. The initial session with one of the investigators will be an introduction and a review of Module 1: Gratitude, and will last 30-60min. Three follow-up sessions will occur approximately every two weeks and the participants should view the videos before those virtual meetings (Session 2 will review Module II: Mindful Presence; Session 3 will review Module III: Kindness; Session 4 will review Module IV: Resilient Mindset). The videos will take approximately 30 minutes each to review and virtual sessions will each take 30-60 minutes.

SUMMARY:
Researchers are trying to find out if the Resilient Living Program will improve quality of life, stress, anxiety, sleep, fatigue, and resilience in patients with advanced cancer and their caregivers.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age ≥18 years
* English fluency
* No diagnosed severe cognitive impairment
* Diagnosis of stage IV solid tumor cancer
* Expected prognosis >6 <18 months
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Patient baseline distress score ≥4/10 OR identified as having distress that would benefit from program by care team or provider
* Ability to do first Resilient Living session in person

Inclusion Criteria for caregivers:

* Self-identifies as a caregiver of a patient that meets the above cancer diagnosis criteria, and who also participates in the study
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Age ≥18 years
* English fluency
* No diagnosed severe cognitive impairment
* Ability to do first Resilient Living session in person

Exclusion Criteria:

* As determined through self-report, those diagnosed with a history of a psychotic episode will be excluded.
* Other psychological co-morbidities such as untreated schizophrenia, bipolar disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress | Baseline; Week 5 (after 2nd session); Week 9 (after 4th session); Week 12 (one month after completing all sessions)
  Stress, as measured by the Perceived Stress Scale (PSS). The PSS has 14 items, 7 positively stated and 7 negatively stated. Likert-type 5-point scale. Positively stated items reverse coded; scores are summed; scores range 0-56. High score indicates greater stress level.
Change in Anxiety | Baseline; Week 5 (after 2nd session); Week 9 (after 4th session); Week 12 (one month after completing all sessions)
  Anxiety, as measured by the Generalized Anxiety Disorder 7-item scale (GAD-7). The GAD-7 has 7 items, about which the participant has felt bothered by in the prior two weeks. 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day. Scores are summed; range 0-21. Score 0-4 minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre R. Pachman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials